CLINICAL TRIAL: NCT01962935
Title: A Phase I Study in Healthy Volunteers to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD4721 After Once Daily Administration of Multiple Ascending Doses for 10 Days, and an Open-label Comparison With the Pharmacodynamics of AZD5069 Given Twice Daily for 3 Days
Brief Title: Study to Investigate Safety, Tolerability and Effect of Multiple Dosing With AZD 4721 and/or With AZD 5069
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D5200C00002
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD).
Keywords: Healthy volunteer; Multiple ascending dose
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — N-(2-(2,3-difluoro-6-benzylthio)-6-(3,4-dihydroxybutan-2-yloxy)pyrimidin-4-yl)azetidine-1-sulfonamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A AZD4721 (Experimental): Part A of the study, multiple ascending doses of AZD4721 will be administrated once daily for 10 days
  Interventions: Drug: AZD4721
- Placebo (Placebo Comparator): Part A of the study, multiple ascending doses of matching Placebo will be administrated once a daily for 14 days
  Interventions: Drug: Placebo
- AZD5069, then AZD4721 (Active Comparator): Part B of the study, subject will participate in two treatment periods (one with AZD5069 administrated for 3 days and the second period with AZD4721 administrated for 14 days) separated by a wash-out period of 6-10 days between the two periods.
  Interventions: Drug: AZD4721; Drug: AZD5069

INTERVENTIONS:
Drug: AZD4721 — Part A - multiple ascending dose, daily; Part B - one dose decided after part A, daily
  Arms: AZD5069, then AZD4721; Part A AZD4721
Drug: Placebo — Part A - multiple ascending dose daily
  Arms: Placebo
Drug: AZD5069 — Part B - one dose decided after part A, twice a day
  Arms: AZD5069, then AZD4721

SUMMARY:
Study to investigate safety, tolerability and effect of multiple dosing with AZD 4721 and/or with AZD 5069

DETAILED DESCRIPTION:
The purpose of the study is to investigate the safety and tolerability, pharmacokinetics and pharmacodynamics of AZD 4721 in healthy volunteers after once daily administration of multiple ascending doses for 10 days, and an open-label comparison with the pharmacodynamics of AZD5069 given twice daily for 3 days

ELIGIBILITY:
Inclusion Criteria:

* 1.Provision of signed and dated, written informed consent prior to any study specific procedures.
* 2.Healthy male and/or female Caucasian (neither Black/African American nor Japanese) volunteers aged 18 to 50 years with suitable veins for cannulation or repeated venipuncture. ("Healthy" is as determined by medical history and physical examination, clinical laboratory parameters, and ECG and performed before first dose administration.).
* 3.Healthy volunteers should have a body mass index (BMI) between 18 and 30 kg/m2 (inclusive) and weigh at least 50 kg and no more than 100 kg (inclusive).

Exclusion Criteria:

1. Pyrexial with a body temperature higher than 37.7°C at Day -1 (Visit 2), or as judged by the investigator.
2. Screening blood neutrophil counts (taken in the morning) not within the laboratory reference range (Visit 1).
3. Other latent or chronic infections (eg, recurrent sinusitis, genital or ocular herpes, urinary tract infection) or at risk of infection (surgery, trauma, or significant infection) in the previous 90 days, or history of skin abscesses within the previous 90 days.
4. Clinically significant lower respiratory tract infection not resolved within 4 weeks prior to screening (Visit 1), as determined by the investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Description of the safety profile in terms of Adverse events; blood pressure, heart rate and body temperature; electrocardiograms; clinical chemistry; haematology assessments | From Admission day -1 up to Follow up ( Max 12 weeks)
  Same for both part A and B
Description of neutrophils in terms of absolute blood neutrophil count ratio [ANC ratio], time of ANCmin,ss [ANCtmin,ss], | Samples taken for part A day -1, Day 1 at predose,1h,2h,6h and 12h postdose, predose day 2,3,4,5,6,7,8,9,10 predose and at 1h,2h,3h,6h,9h,12h,15h,18h,21h,24h,36h,48h post last dose ( given day 10).
  Part A AZD4721
Description of neutrophils in terms of minimum ANC during first 24 hours on Day 1 [Part A only, ANCmin,Day 1], time of ANCmin,Day 1 [ANCtmin,Day 1], minimum ANC ratio during first 24 hours on Day 1 [Part A only, ANCmin ratio,Day 1] | Samples taken for Part A Day 1 at predose, 1h,2h,6h12h and 24h postdose.
  Part A AZD4721
Descriptions of neutrophils in terms of minimum ANC during the 24 hours following the last morning dose [ANCmin,ss], mean of ANC values during the 24 hours following the last morning dose [ANCmean,ss], | Samples taken for Part A day10 predose and at 1h,2h,3h,6h,9h,12h,15h,18h,21h,24h post dose
  Part A AZD4721
Description of neutrophils in terms of minimum ANC ratio during the 24 hours following the last morning dose [ANCmin ratio,ss], and mean of ANC ratio values during the 24 hours following the last morning dose [ANCmean ratio,ss]). | Samples taken for Part A day 10 predose and at 1h,2h,3h,6h,9h,12h,15h,18h,21h,24h post dose
  Part A AZD4721
Description of neutrophils in terms of • absolute blood neutrophil count ratio [ANC ratio], time of ANCmin,ss [ANCtmin,ss], | Part B visit 1 day -1, day 1 predose, 12h, day 2 predose, day 3 predose,3h,6h,9h,12h,15h,18h,21h and 24h post dose
  Part B AZD5069
Description of neutrophils in terms of • time of ANCmin,Day 1 [ANCtmin,Day 1], | Part B day 1 predose, 12h and 24h postdose
  Part B AZD5069
Description of neutrophile in terms of minimum ANC during the 24 hours following the last morning dose [ANCmin,ss], mean of ANC values during the 24 hours following the last morning dose [ANCmean,ss] | Samples taken Part B day 3 predose,3h,6h,9h,12h,15h,18h,21h and 24h post dose
  Part B AZD5069
Description of neutrophils in terms of minimum ANC ratio during the 24 hours following the last morning dose [ANCmin ratio,ss], and mean of ANC ratio values during the 24 hours following the last morning dose [ANCmean ratio,ss]). | Samples taken Part B day 3 predose,3h,6h,9h,12h,15h,18h,21h and 24h post dose
  Part B AZD5069
Description of neutrophils in terms of • absolute blood neutrophil count ratio [ANC ratio], time of ANCmin,ss [ANCtmin,ss] | Samples taken for part B day -1, predose day 1,2,4,6,8,10 and at 1h,2h,3h,6h,9h,12h,15h,18h,21h,24h post dose
  Part B AZD4721
Description of neutrophils in terms of time of ANCmin,Day 1 [ANCtmin,Day 1], | Samples taken for part B predose day 1
  Part B AZD4721
Description of neutrophils in terms of minimum ANC during the 24 hours following the last morning dose [ANCmin,ss], mean of ANC values during the 24 hours following the last morning dose [ANCmean,ss] | Samples taken part B pre dose day 10 and at 1h,2h,3h,6h,9h,12h,15h,18h,21h,24h post dose
  Part B AZD4721
Description of neutrophils in terms of minimum ANC ratio during the 24 hours following the last morning dose [ANCmin ratio,ss], and mean of ANC ratio values during the 24 hours following the last morning dose [ANCmean ratio,ss]). | Samples taken part B pre dose day 10 and at 1h,2h,3h,6h,9h,12h,15h,18h,21h,24h post dose
  Part B AZD4721

SECONDARY OUTCOMES:
Description of the pharmacokinetic(PK) profile of AZD 4721 in terms of Maximum plasma concentration (Cmax), maximum plasma concentration divided by dose (Cmax/D), time to Cmax (tmax) | Sample taken Day 1 post dose at 0:20, 0:40,1h, 2h,3h,6h,9h,12h,15h,18h,21h and 24h.
  Following single dose administration of AZD4721 Part A
Description of the PK profile of AZD 4721 in terms of area under the plasma concentration-time curve during the dosing interval (AUCtau),), lag-time (tlag), ratio of metabolite AUCtau to parent AUCtau (MRAUC) | Sample taken Day 1 post dose at 0:20, 0:40,1h, 2h,3h,6h,9h,12h,15h,18h,21h and 24h.
  Following single dose administration of AZD4721 Part A
Description of the PK profile of AZD 4721 in terms of ratio of metabolite Cmax to parent Cmax (MRCmax) | Sample taken Day 1 post dose at 0:20, 0:40,1h, 2h,3h,6h,9h,12h,15h,18h,21h and 24h.
  Following single dose administration of AZD4721 Part A
Description of the PK profile of AZD 4721 in terms of Maximum plasma concentration (Css,max), maximum plasma concentration divided by dose (Css,max/D) time to Css,max (tss,max) | Sample taken Day 1 post dose at 0:20, 0:40,1h, 2h,3h,6h,9h,12h,15h,18h,21h and 24h. Predose day 3,4,5,6,7,8,9,10 and at 0:20,0:40,1h,2h,3h,6h,9h,12h,15h,18h,21h,24h,48h,72h and 96h post last dose
  Following multiple dose administration of AZD4721Part A
Description of the PK profile of AZD 4721 in terms of minimum plasma concentration (Css,min)), time to Css,min (tss,min) average concentration over the investigational product interval (Css,av) | Sample taken Day 1 post dose at 0:20, 0:40,1h, 2h,3h,6h,9h,12h,15h,18h,21h and 24h. Predose day 3,4,5,6,7,8,9,10 and at 0:20,0:40,1h,2h,3h,6h,9h,12h,15h,18h,21h,24h,48h,72h and 96h post last dose
  Following multiple dose administration of AZD4721 Part A
Description of the PK profile of AZD 4721 in terms of peak to trough concentration ratio (Css,max/Css,min)), terminal rate constant (z), terminal half-life (t1/2λz) | Sample taken Day 1 post dose at 0:20, 0:40,1h, 2h,3h,6h,9h,12h,15h,18h,21h and 24h. Predose day 3,4,5,6,7,8,9,10 and at 0:20,0:40,1h,2h,3h,6h,9h,12h,15h,18h,21h,24h,48h,72h and 96h post last dose
  Following multiple dose administration of AZD4721 Part A
Description of the PK profile of AZD 4721 in terms of area under the plasma concentration-time curve during the dosing interval at steady state (AUCss,tau), AUCss,tau divided by dose (AUCss,tau/D) | Sample taken Day 1 post dose at 0:20, 0:40,1h, 2h,3h,6h,9h,12h,15h,18h,21h and 24h. Predose day 3,4,5,6,7,8,9,10 and at 0:20,0:40,1h,2h,3h,6h,9h,12h,15h,18h,21h,24h,48h,72h and 96h post last dose
  Following multiple dose administration of AZD4721Part A
Description of the PK profile of AZD 4721 in terms of apparent clearance (CL/F), ), volume of distribution (Vz/F) | Sample taken Day 1 post dose at 0:20, 0:40,1h, 2h,3h,6h,9h,12h,15h,18h,21h and 24h. Predose day 3,4,5,6,7,8,9,10 and at 0:20,0:40,1h,2h,3h,6h,9h,12h,15h,18h,21h,24h,48h,72h and 96h post last dose
  Following multiple dose administration of AZD4721 Part A
Description of the PK profile of AZD 4721 and metabolite in terms of ratio of metabolite AUCss,tau to parent AUCss,tau (MRAUCss,tau), ratio of metabolite Css,max to parent Css,max (MRCss,max) | Sample taken Day 1 post dose at 0:20, 0:40,1h, 2h,3h,6h,9h,12h,15h,18h,21h and 24h. Predose day 3,4,5,6,7,8,9,10 and at 0:20,0:40,1h,2h,3h,6h,9h,12h,15h,18h,21h,24h,48h,72h and 96h post last dose
  Following multiple dose administration of AZD4721 Part A
Description of the PK profile of AZD 4721 and metabolite in terms of accumulation ratio for AUCtau (RAUCtau), and accumulation ratio for Cmax (RCmax). | Sample taken Day 1 post dose at 0:20, 0:40,1h, 2h,3h,6h,9h,12h,15h,18h,21h and 24h. Predose day 3,4,5,6,7,8,9,10 and at 0:20,0:40,1h,2h,3h,6h,9h,12h,15h,18h,21h,24h,48h,72h and 96h post last dose
  Following multiple dose administration of AZD4721 Part A
Description of the PK profile of AZD 4721 in terms of Cumulative amount of AZD4721 and AZ13622093 excreted over the investigational product administration interval (Ae (0-tau)) | Urine collection 24h from 0h-24 day 10
  Following multiple dose administration of AZD4721 Part A
Description of the PK profile of AZD 4721 in terms of fraction of dose excreted into the urine over the dosing interval for AZD4721 (fe (0 tau)), and renal clearance (CLR). | Urine collection 24h from 0h-24 day 10
  Following multiple dose administration of AZD4721 Part A
Description of PK Profile of AZD5069 in terms of observed global maximum concentration (Css,max), time to global Css,max (tss,max), observed global minimum concentration (Css,min) | Sample taken day 1 12h, day 2 0h and 12h, day 3 0h,3h,6h,9h,12h,15h,18h,21h and 24h post dose
  Following multiple dosing of AZD5069 Part B
Description of PK Profile of AZD5069 in terms of time to global Css,min (tss,min), average concentration over 24 hours (Css,av), peak to trough concentration ratio (Css,max/Css,min) | Sample taken day 1 12h, day 2 0h and 12h, day 3 0h,3h,6h,9h,12h,15h,18h,21h and 24h post dose
  Following multiple dosing of AZD5069 Part B
Description of PK Profile of AZD5069 in terms of AUC during the 12 hour interval after the morning dose(AUCtau,morning), AUC during the 12 hour dosing interval after the evening dose (AUCtau,evening) | Sample taken day 1 12h, day 2 0h and 12h, day 3 0h,3h,6h,9h,12h,15h,18h,21h and 24h post dose
  Following multiple dosing of AZD5069 Part B
Description of PK Profile of AZD5069 in terms of and area under the plasma concentration time curve 0 to 24 hours post morning dose (AUC(0 24h)). | Sample taken day 1 12h, day 2 0h and 12h, day 3 0h,3h,6h,9h,12h,15h,18h,21h and 24h post dose
  Following multiple dosing of AZD5069 Part B
Description of PK Profile of AZD4721 in terms of maximum plasma concentration (Css,max), time to Css,max (tss,max), minimum plasma concentration (Css,min), time to Css,min (tss,min), average concentration over the dosing interval (Css,av) | Sample taken predose Day 2,4,6,8,10 and at 0:20h,0:40h,1h,2h,3h,6h,9h,12h,15h,18h,21h and 24h post dose
  Following multiple dosing of AZD4721 Part B
Description of PK Profile of AZD4721 in terms of peak to trough concentration ratio (Css,max/Css,min), area under the plasma concentration time curve during the dosing interval (AUCss,tau), and apparent clearance (CL/F). | Sample taken predose Day 2,4,6,8,10 and at 0:20h,0:40h,1h,2h,3h,6h,9h,12h,15h,18h,21h and 24h post dose
  Following multiple dosing of AZD4721 Part B

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Siew, MD, Principal Investigator — Quintiles London, UK; Bengt Larsson, MD, Study Director — Astrazeneca Mölndal, Sweden
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1878&filename=D5200C00002_Study_Synopsis.pdf